CLINICAL TRIAL: NCT06003413
Title: Evaluation of the Relationship Between the Architecture of the Quadriceps, Tibialis Anterior and Gastrocnemius Muscles and Muscle Strength in Female Gonarthrosis Patients
Brief Title: Evaluation of the Relationship Between Muscle Architecture and Muscle Strength in Female Gonarthrosis Patients
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/162
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Osteo Arthritis Knee; Gonarthrosis; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Osteoarthritic Knee: * Knees with Kellgren-Lawrence Stage 2-4 will admitted to this group
  * Vastus Lateralis, Tibialis Anterior, Lateral Gastrocnemius and Medial Gastrocnemius ultrasonography will be performed to evaluate muscle thickness, pennation angle and fascicle length.
  * Outcome Measures in Rheumatology (OMERACT) Ultrasound scores for knee will be evaluated
  * Isometric knee extension, isometric ankle dorsiflexion and isometric ankle plantar flexion strength will be evaluated with hand held dynamometer
- Healthy Knee: * Healthy knees will be admitted to this group
  * Vastus Lateralis, Tibialis Anterior, Lateral Gastrocnemius and Medial Gastrocnemius ultrasonography will be performed to evaluate muscle thickness, pennation angle and fascicle length.
  * Isometric knee extension, isometric ankle dorsiflexion and isometric ankle plantar flexion strength will be evaluated with hand held dynamometer

SUMMARY:
The goal of this cross-sectional study is to evaluate muscle architecture changes and it's effect on muscle strength in female patients with gonarthrosis.Main questions are:

* Is there any correlation between muscle strength and muscle thickness, pennation angle fiber length?
* Is there any muscle architecture difference in gonarthrosis and is it effecting the muscle strength? The investigators will enroll patients with unilateral gonarthrosis so that investigators can compare the changes within osteoarthritic and healthy knee with the same physical activity levels.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a chronic disease characterized by morning stiffness, reduced joint range of motion, chronic pain, and decreased muscle strength, leading to functional limitations as the disease progresses . In patients with knee osteoarthritis, all muscles of the hip, knee, and ankle are affected in some way . Evidence suggests that impairments in muscle strength in the lower extremities contribute to increased pain and joint space narrowing. Voluntary muscle contractions lead to various changes in muscle architecture, including changes in fascicle angle and pennation angle as well as muscle thickness. While muscle cross-sectional area and thickness are primarily associated with the magnitude of generated force, parameters such as pennation angle have been found to be more related to explosive force. Ultrasonography (US) is a non-invasive imaging method that can visualize these changes. Muscle architecture parameters obtained from US can provide reliable data related to muscle contractility independently of surrounding muscles. Furthermore, US is considered to have similar validity to MRI imaging, which is the gold standard for displaying muscle architecture. Additionally, isometric muscle strength can be reliably measured using handheld dynamometers. Although studies have investigated the relationship between muscle strength and muscle architecture determined by US in patients with knee OA, these studies have predominantly examined the relationship in the quadriceps muscle, and muscles associated with the ankle have not been studied extensively.

ELIGIBILITY:
Inclusion Criteria:

* To be ≥18 years of age,
* Presence of unilateral knee OA (according to American College of Rheumatology criteria),
* Presence of knee OA with Kellgren/Lawrence (K/L) stage ≥2,
* Ability to live independently,
* Ability to walk without assistive devices.

Exclusion Criteria:

* History of surgery on the spine or lower extremities,
* History of inflammatory rheumatic disease,
* Severe cardiovascular disease,
* Neuromuscular disease affecting muscle strength,
* Individuals following a regular exercise program,
* Secondary osteoarthritis.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients who applied to the Bezmialem Vakıf University, Physical Medicine and Rehabilitation Outpatient Clinic appropriate for eligibility criteria will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | 1 day
  Self reported pain scored between 0 (minimum)-10 (maximum). Higher scores represent a worse outcome.
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 1 day
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) was created to assess pain, stiffness, and physical function in patients with hip and / or knee osteoarthritis (OA).
  The WOMAC consists of 24 items divided into 3 subscales:
  * Pain (5 items):
  * Stiffness (2 items):
  * Physical Function (17 items) Number of items in scale: 24 items The WOMAC is available in 5-point Likert-type and 100mm Visual Analog formats
Isometric Knee Extension Muscle Strength | 1 day
  Isometric Knee Extension Muscle Strength will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.
Isometric Ankle Dorsiflexion Muscle Strength | 1 day
  Isometric Ankle Dorsiflexion Muscle Strength will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.
Isometric Ankle Plantar Flexion Muscle Strength | 1 day
  Isometric Ankle Plantar Flexion Muscle Strength will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.
Health Assessment Questionnaire (HAQ) | 1 day
  The Health assessment questionnaire (HAQ) is a questionnaire for the assessment of disability in an individual. The patients report the amount of difficulty they have in performing eight daily living activities. Each question asks on a scale ranging from 0 to 3 if the categories can be performed without any difficulty (scale 0) up to cannot be done at all (scale 3). The final score varies between 0 and 3.
Outcome Measures in Rheumatology (OMERACT) ultrasound scores for knee osteoarthritis (OA) | 1 day
  The US scores for 7 disease manifestations were then graded by the same operator using the OMERACT knee US OA atlas: semiquantitative scores for (1) synovitis (0-3; combined synovial hypertrophy and effusion); (2) binary scores (0-1) for synovial hypertrophy ≥ 4 mm, (3) effusion ≥ 4 mm12; and (4) Power Doppler (PD) signals separate from suprapatellar recess in a longitudinal plane, medial and lateral parapatellar recesses in a transverse plane, semiquantitative scores for (5) osteophytes (0-3) from the medial and lateral joint aspects in a longitudinal plane and (6) meniscal extrusion (0-2; only the medial joint aspects) in a longitudinal plane, and for (7) cartilage abnormalities (0-3) in a transverse plane on a maximally flexed knee

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Volkan Yurdakul, Assoc. Prof., Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Michael JW, Schluter-Brust KU, Eysel P. The epidemiology, etiology, diagnosis, and treatment of osteoarthritis of the knee. Dtsch Arztebl Int. 2010 Mar;107(9):152-62. doi: 10.3238/arztebl.2010.0152. Epub 2010 Mar 5. PMID 20305774
- [Background] Varbakken K, Loras H, Nilsson KG, Engdal M, Stensdotter AK. Relative difference in muscle strength between patients with knee osteoarthritis and healthy controls when tested bilaterally and joint-inclusive: an exploratory cross-sectional study. BMC Musculoskelet Disord. 2019 Dec 9;20(1):593. doi: 10.1186/s12891-019-2957-6. PMID 31818286
- [Background] Glass NA, Torner JC, Frey Law LA, Wang K, Yang T, Nevitt MC, Felson DT, Lewis CE, Segal NA. The relationship between quadriceps muscle weakness and worsening of knee pain in the MOST cohort: a 5-year longitudinal study. Osteoarthritis Cartilage. 2013 Sep;21(9):1154-9. doi: 10.1016/j.joca.2013.05.016. PMID 23973125
- [Background] Fukunaga T, Ichinose Y, Ito M, Kawakami Y, Fukashiro S. Determination of fascicle length and pennation in a contracting human muscle in vivo. J Appl Physiol (1985). 1997 Jan;82(1):354-8. doi: 10.1152/jappl.1997.82.1.354. PMID 9029238
- [Background] Hodges PW, Pengel LH, Herbert RD, Gandevia SC. Measurement of muscle contraction with ultrasound imaging. Muscle Nerve. 2003 Jun;27(6):682-92. doi: 10.1002/mus.10375. PMID 12766979
- [Background] Bazyler CD, Mizuguchi S, Harrison AP, Sato K, Kavanaugh AA, DeWeese BH, Stone MH. Changes in Muscle Architecture, Explosive Ability, and Track and Field Throwing Performance Throughout a Competitive Season and After a Taper. J Strength Cond Res. 2017 Oct;31(10):2785-2793. doi: 10.1519/JSC.0000000000001619. PMID 27575250
- [Background] Gerstner GR, Thompson BJ, Rosenberg JG, Sobolewski EJ, Scharville MJ, Ryan ED. Neural and Muscular Contributions to the Age-Related Reductions in Rapid Strength. Med Sci Sports Exerc. 2017 Jul;49(7):1331-1339. doi: 10.1249/MSS.0000000000001231. PMID 28166121
- [Background] Zaras ND, Stasinaki AN, Methenitis SK, Krase AA, Karampatsos GP, Georgiadis GV, Spengos KM, Terzis GD. Rate of Force Development, Muscle Architecture, and Performance in Young Competitive Track and Field Throwers. J Strength Cond Res. 2016 Jan;30(1):81-92. doi: 10.1519/JSC.0000000000001048. PMID 26049793
- [Background] Zhang Q, Sheng Z, Moore-Clingenpeel F, Kim K, Sharma N. Ankle Dorsiflexion Strength Monitoring by Combining Sonomyography and Electromyography. IEEE Int Conf Rehabil Robot. 2019 Jun;2019:240-245. doi: 10.1109/ICORR.2019.8779530. PMID 31374636
- [Background] Walton JM, Roberts N, Whitehouse GH. Measurement of the quadriceps femoris muscle using magnetic resonance and ultrasound imaging. Br J Sports Med. 1997 Mar;31(1):59-64. doi: 10.1136/bjsm.31.1.59. PMID 9132215
- [Background] Wang CY, Olson SL, Protas EJ. Test-retest strength reliability: hand-held dynamometry in community-dwelling elderly fallers. Arch Phys Med Rehabil. 2002 Jun;83(6):811-5. doi: 10.1053/apmr.2002.32743. PMID 12048660
- [Background] Malas FU, Ozcakar L, Kaymak B, Ulasli A, Guner S, Kara M, Akinci A. Effects of different strength training on muscle architecture: clinical and ultrasonographic evaluation in knee osteoarthritis. PM R. 2013 Aug;5(8):655-62. doi: 10.1016/j.pmrj.2013.03.005. Epub 2013 Mar 7. PMID 23474211
- [Background] Blazevich AJ, Cannavan D, Coleman DR, Horne S. Influence of concentric and eccentric resistance training on architectural adaptation in human quadriceps muscles. J Appl Physiol (1985). 2007 Nov;103(5):1565-75. doi: 10.1152/japplphysiol.00578.2007. Epub 2007 Aug 23. PMID 17717119
- [Background] Taniguchi M, Fukumoto Y, Kobayashi M, Kawasaki T, Maegawa S, Ibuki S, Ichihashi N. Quantity and Quality of the Lower Extremity Muscles in Women with Knee Osteoarthritis. Ultrasound Med Biol. 2015 Oct;41(10):2567-74. doi: 10.1016/j.ultrasmedbio.2015.05.014. Epub 2015 Jun 20. PMID 26099784